CLINICAL TRIAL: NCT06689254
Title: REVERSE: a Randomized Controlled Trial (RCT) to Ameliorate Treatment-resistant Post Traumatic Stress Disorder (PTSD) with Glucocorticoid Receptor (GR) Antagonism
Brief Title: REVERSE: Improving Treatment-resistant Post Traumatic Stress Disorder (PTSD) with Glucocorticoid Receptor (GR) Antagonism
Acronym: REVERSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christiaan Vinkers (Other)
Collaborators: Corcept Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Christiaan Vinkers, Prof., Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REVERSE; 2024-511042-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-29; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Treatment-resistant PTSD
Keywords: PTSD; GR-antagonism; mifepristone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mifepristone (Experimental)
  Interventions: Drug: Mifepristone 1200 mg daily
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone 1200 mg daily — Oral tablets
  Arms: Mifepristone
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
Rationale:

Post-traumatic stress disorder (PTSD) is a psychiatric disorder that can develop in people who have experienced or witnessed a traumatic event. Symptoms of PTSD include flashbacks, nightmares, difficulty sleeping, difficulty concentrating, irritability, and avoidance of people, places, or activities that remind the person of the traumatic event. Even though there are effective treatments (e.g. exposure-based psychotherapies and antidepressants), not all patients respond. Glucocorticoid receptor (GR) antagonism is a potential therapy for the treatment of treatment-resistant post traumatic stress disorder (PTSD) based on the idea that PTSD may be caused or exacerbated by dysregulation of the body's stress response system, and on the results of several small clinical trials. By blocking the actions of cortisol at the GR, it is thought that GR antagonists may be able to reduce the severity of PTSD symptoms and improve treatment outcomes. Randomized controlled trials (RCT) can provide high-quality evidence on treatment efficacy, and optimize evidence-based selection of off-label treatments for patients. Therefore the aim is to investigate whether the psychological and biological sequelae of traumatic stress and PTSD can be targeted by blocking the glucocorticoid receptor (GR) using the generic drug mifepristone in a double blind, placebo controlled RCT.

Objective:

To test the hypothesis that treatment with the GR-antagonist mifepristone is more effective than placebo to reduce PTSD symptom severity in treatment-resistant PTSD.

Main trial endpoints:

Improvement of PTSD symptoms, as measured with the monthly version of the CAPS-5 (Clinician Administered PTSD scale) in patients with treatment-resistant PTSD, 4 weeks after the start of the intervention. Secondary trial endpoints

* PTSD symptom severity as measured with the weekly version of the PCL-5, from baseline till 12 weeks after the start of the intervention (T3).
* Long-term PTSD symptom severity as measured with the CAPS-5, at 12 weeks after the start of the intervention (T3).
* Loss of diagnosis (score of <26 and absence of PTSD criteria with CAPS-5), 4 weeks after the start of the intervention.
* Treatment response (minimum decrease of 10 point on the PCL-5 and CAPS-5 scores) at 1, 4 and 12 weeks after the start of the intervention.
* Other clinical outcomes 1, 4, and 12 weeks after the start the intervention:

  * disability (WHO Disability Schedule 2.0; WHO-DAS II),
  * sleep (Insomnia Severity Index; ISI),
  * subjective stress (Perceived Stress Scale; PSS),
  * anxiety symptoms (Beck Anxiety Inventory; BAI),
  * depressive symptoms (IDS-SR),
  * suicidal ideation and behaviour (Columbia-Suicide Severity Rating Scale).

Trial design:

The experimental protocol consists of a placebo-controlled double-blind RCT with 4 face-to-face meetings:

* baseline (T0, 2,5 hrs);
* post-intervention T1, 8 days after start (1hr);
* post-intervention T2, 4 weeks after start (2hr).
* post-intervention T3, 12 weeks (2hr).

Trial population:

60 adult patients (male/female, 18+ years), with treatment-resistant PTSD (non-response to two evidence-based PTSD treatments, at least one of which is trauma-focused psychotherapy). Intervention Patients are randomized for treatment with the GR antagonist mifepristone (1200 mg/day for 7 days) or matching placebo (daily for 7 days). Study medication will be dispensed during the baseline measurement (T0), and taken once daily for 7 consecutive days. Clinical measurements consist of clinical interviews and questionnaires. During baseline visits a pregnancy test is conducted in woman of child bearing potential (WOCBP), and blood is drawn at T1 to assess mifepristone plasma levels.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks:

Mifepristone has been clinically used for Cushing's syndrome (anti-glucocorticoid effects) and termination of pregnancy (anti-progesterone effects) for several decades. Mifepristone is generally well-tolerated, and several double-blind studies using the identical duration and dose have shown (7 days, 1200 mg) that the safety profile of mifepristone is comparable to that of placebo treatment, and study dropouts due to side effects were higher for placebo (1.6%) than for mifepristone (1.4%). The most common adverse events (AEs) were nausea, headache, dizziness, and a dry mouth and were comparable between the mifepristone and placebo groups. With regard to mifepristone's progesterone receptor activity and its indication for pregnancy termination, WOCBP who do not agree to use a non-hormonal contraceptive method (condom) during the intervention and up to 1 month after the intervention, are strictly excluded from participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Mastery of Dutch language
* Age of ≥ 18 years of age and able to give written IC
* Participant agrees to be randomized
* DSM-5 diagnosis of PTSD, confirmed with clinical interview (CAPS-5)
* Treatment-resistant PTSD

  * CAPS-5 score ≥ 30
  * Nonresponse to two evidence-based treatments for PTSD recommended by a recent clinical practice guidelines delivered with fidelity and at an effective dose, at least one of which is a full course of trauma-focused psychotherapy

Exclusion Criteria:

* Bipolar disorder, psychotic disorder, or current alcohol/drug dependence that requires clinical attention.
* Female participant being a WOCBP and who does not want to use a non-hormonal contraceptive method (condom) during the intervention period and up to 1 month after the intervention.
* Female participants that are pregnant or breastfeeding. Pregnancy is excluded using a negative highly sensitive pregnancy test before the first dose of the study medication during the baseline visit.
* Female participants that have a history of unexplained vaginal bleeding or endometrial changes.
* Chronic adrenal insufficiency.
* Current use of:

  * Medications containing CYP3A4-inhibitors, as an interaction of CYP3A4-inhibitors and mifepristone leads to higher mifepristone plasma levels and increases the chance of having side effects. This also includes the consumption of grapefruit juice during the intervention
  * Medications containing CYP3A4-inductors, as an interaction of CYP3A4-inductors and mifepristone leads to lower mifepristone plasma levels and decreases the chance of having a beneficial effect. This also includes the consumption of St John's worth/hypericum perforatum during the intervention.
  * Medications containing CYP3A4 substrates.
  * Medications containing CYP2C8/9 substrates.
  * Medications containing P-gp and BCRP transported drugs
  * Glucocorticoid antagonists within 1 week before possible start of trial treatment.
  * Systemic corticosteroids. Topical corticosteroid treatment are acceptable, with the exception of inhaled corticosteroids (inhalators).
  * Unstable drug dosages (e.g. tapering of antidepressants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Improvement of PTSD symptoms | 4 weeks after the start of the intervention (T2)
  Measured with the monthly version of the CAPS-5 (Clinician Administered PTSD scale) in patients with treatment-resistant PTSD. Minimum and maximum score range from 0-80, with higher scores indicating greater PTSD symptom severity.

SECONDARY OUTCOMES:
PTSD symptom severity | From baseline till 12 weeks after the start of the intervention (T3)
  Measured with the weekly version of the PTSD checklist for the DSM-5 (PCL-5). Minimum and maximum score range from 0-80, with higher scores indicating greater PTSD symptom severity.
Long-term PTSD symptom severity | 12 weeks after the start of the intervention (T3)
  Measured with the Clinician Administered PTSD scale (CAPS-5). Minimum and maximum score range from 0-80, with higher scores indicating greater PTSD symptom severity.
Loss of diagnosis | 4 weeks after the start of the intervention (T2)
  Score of <26 and absence of PTSD criteria on the Clinician Administered PTSD scale (CAPS-5). Dichotomous outcome with yes/no loss of diagnosis. Minimum and maximum score range from 0-80, with higher scores indicating greater PTSD symptom severity.
Treatment response | 1, 4 and 12 weeks after the start of the intervention (T1, T2, T3)
  Minimum decrease of 10 point on the Clinician Administered PTSD scale (CAPS-5). Dichotomous outcome indicating loss of diagnosis (yes/no). Minimum and maximum score range from 0-80, with higher scores indicating greater PTSD symptom severity.
Treatment response | 1, 4 and 12 weeks after the start of the intervention (T1, T2, T3)
  Minimum decrease of 10 point on the PTSD checklist for the DSM-5 (PCL-5). Dichotomous outcome indicating loss of diagnosis (yes/no). Minimum and maximum score range from 0-80, with higher scores indicating greater PTSD symptom severity.
Disability | 1, 4, and 12 weeks after the start the intervention (T1, T2, T3)
  WHO Disability Schedule 2.0; WHO-DAS II. Minimum and maximum score range from 0-100, with higher scores indicating greater severity.
Sleep | 1, 4, and 12 weeks after the start the intervention ( T1, T2, T3)
  Insomnia Severity Index; ISI. Minimum and maximum score range from 0-28, with higher scores indicating greater severity.
Subjective stress | 1, 4, and 12 weeks after the start the intervention (T1, T2, T3)
  Perceived Stress Scale; PSS. Minimum and maximum score range from 0-40, with higher scores indicating greater severity.
Anxiety symptoms | 1, 4, and 12 weeks after the start the intervention (T1, T2, T3)
  Beck Anxiety Inventory; BAI. Minimum and maximum score range from 0-63, with higher scores indicating greater severity.
Depressive symptoms | 1, 4, and 12 weeks after the start the intervention (T1, T2, T3)
  Inventory of Depressive Symptomatology Self Report; IDS-SR. Minimum and maximum score range from 0-84, with higher scores indicating greater severity.
Suicidal ideation and behaviour | 1, 4, and 12 weeks after the start the intervention (T1, T2, T3)
  Columbia-Suicide Severity Rating Scale; C-SSRS. Minum to maximum score range from 0-25, with higher scores indicating greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided